CLINICAL TRIAL: NCT02014896
Title: Ischemia Care Biomarkers of Acute Stroke Etiology (BASE)
Acronym: BASE
Status: Completed | Type: Observational
Sponsor: Ischemia Care LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ISCH01
Record Dates: First submitted 2013-12-05; First posted 2013-12-18 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Ischemic Stroke; Atrial Fibrillation; Transient Ischemic Attacks; Transient Cerebrovascular Events; Thrombotic Stroke; Stroke of Basilar Artery; Cardioembolic Stroke
Keywords: Ischemic Stroke; Transient Ischemic Attack; Transient Neurological Event; Atrial Fibrillation; Cryptogenic Stroke; Gene Expression; RNA; Anticoagulant; NOAC; Antiplatelet; Cardiac monitoring; Point of Care; tPA; Atheroembolic
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Ischemic Attack, Transient; Thrombotic Stroke; Embolic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen will be whole blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Ischemic Stroke: Ischemic stroke subjects presenting within 24 hours from symptom onset will have serial PAX Gene Blood RNA tubes drawn within 18 hours of onset of symptoms upon arrival to the Emergency Department (if available) or hospital; 24 hours +/- 6 hours from symptom onset (if available) and 48 hours+/- 6 hours from symptom onset (if available).
  Biomarker blood draw
  Interventions: Other: Biomarker blood draw
- TIA (Transient Ischemic Attack): TIA subjects presenting within 24 hours from symptom onset will have serial PAX Gene Blood RNA tubes drawn within 18 hours of onset of symptoms upon arrival to the Emergency Department (if available) or hospital; 24 hours +/- 6 hours from symptom onset (if available) and 48 hours+/- 6 hours from symptom onset (if available).
  Biomarker blood draw
  Interventions: Other: Biomarker blood draw
- Non-Ischemic TNE: Non-Ischemic Transient Neurological Event (TNE) subjects will have serial PAX Gene Blood RNA tubes drawn within 18 hours of onset of symptoms upon arrival to the Emergency Department or hospital.
  Biomarker blood draw
  Interventions: Other: Biomarker blood draw
- Control: Control group subjects will have PAX Gene Blood RNA tubes drawn within 8 hours of arrival to the Emergency Department or hospital. Control group matched with ischemic stroke and TIA subjects for age, race, gender, smoking history with at least one of the following vascular risk factors: diabetes, hypertension, atrial fibrillation, hyperlipidemia.
  Biomarker blood draw
  Interventions: Other: Biomarker blood draw

INTERVENTIONS:
Other: Biomarker blood draw — Comparison of gene expression profiles using RNA isolated from whole blood.
  Other Names: PAX Gene Blood RNA tube, PreAnalytiX, Germnay

SUMMARY:
The proposed study will validate the clinical use of new biomarker blood tests to identify blood components that may differentiate between diverse stroke etiologies and clinical outcomes as listed below:

1. Differentiate between cardioembolic and large artery atherosclerotic ischemic strokes, when hemorrhagic stroke is ruled out.
2. In cases of ischemic strokes of unknown or "cryptogenic" etiology, determine the ability of biomarker blood tests to predict etiology between cardioembolic and large artery atherosclerotic.
3. In cases of cardioembolic ischemic stroke, further differentiation of cardioembolic ischemic strokes into those caused by atrial fibrillation (AF) and those not caused by AF.
4. Differentiate "transient ischemic attacks" (TIAs) from acute ischemic strokes.
5. Differentiate TIAs from non-ischemic "transient neurological events" (TNE) with similar symptoms.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a leading cause of adult mortality and morbidity in the United States, affecting over 800,000 individuals, annually, leaving many with permanent disability. Furthermore, hundreds of thousands of Americans experience a transient ischemic attack (TIA), a momentary episode of neurologic dysfunction, which often precedes a major stroke and serves as a warning for future ischemic events. Despite symptoms resolving, experiencing a TIA increases the risk of stroke by 20% within 90 days. Emergent evaluation, prompt acute treatment, and identification of stroke etiology for secondary prevention are key to decreasing the morbidity and mortality associated with cerebrovascular disease. Key to treatment and prevention is the identification of stroke etiology - large vessel atherosclerosis, cardioembolic phenomenon, or in-situ small vessel cerebrovascular disease - since primary and secondary prevention measures differ based on stroke subtype. The diagnosis of ischemic stroke includes a combination of patient history, clinical assessment, and brain imaging. However, identifying the cause of cerebrovascular ischemia is challenging and routinely assigned of cryptogenic origin.

Therefore, there is a great need to understand the pathogenesis of TIA and AIS events in order to develop more effective preventative measures. Recent studies have identified the differential expression of genes in whole blood that may differentiate the major ischemic stroke types. Such differences may help identify TIA and AIS events that are more likely to respond to therapy specifically tailored to the major stroke type. Furthermore, by establishing a more robust standard for secondary prevention, future stroke events may be avoided.

BASE is a multisite prospective study with a estimated enrollment of up to 1100 subjects adult subjects and 100 age, gender and co-morbidity matched controls ("Controls") will be recruited from patients who present to the Emergency Department (ED) or hospital with suspected AIS or TIA. Research personnel will identify potential patients by responding to "Brain Attacks" pages from the ED to the Stroke Team for patients who meet current Brain Attack criteria. Following evaluation by the ED and neurology physicians, the clinical coordinator will verify the patient had a suspected AIS or TIA and meets eligibility criteria. The patient or their legal surrogate will be approached for study participation. Written informed consent will be obtained for all subjects enrolled.

There are two recruitment windows related to BASE determined by time of symptom onset, time of presentation at ED or hospital, and ability to consent:

1. "BASE" - patients that present with suspected stroke symptoms within 18 hours of symptom onset or last known normal time OR
2. "BASE 24" - patients that present within 24 hours +/- 6 hours (i.e. 18 - 30 hour window) of symptom onset or last known normal time and clinical evidence suggesting Acute Ischemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Signs and symptoms suggestive of AIS or TIA
* One of the following:

  1. BASE - Arrival to the emergency department or hospital within 18 hrs of symptom onset or last known normal time
  2. BASE 24 - Arrival to the emergency department or hospital within 24 hours +/- 6 hours (i.e. 18 - 30 hour window) of symptom onset or last known normal time and clinical evidence suggesting Acute Ischemic Stroke.
* Head CT or MRI ruling out other pathology such as vascular malformation, hemorrhage, tumor or abscess which would likely be responsible for presenting neurologic symptoms
* Informed consent obtained

Exclusion Criteria:

* Any central nervous system infection, i.e. meningitis or encephalitis in the past 30 days
* Any form of head trauma, stroke or intracranial hemorrhage in the past 30 days
* Known primary or metastatic cancer involving the brain
* Active Cancer defined as a diagnosis of cancer, within 6 months before enrollment, any treatment for cancer within the previous 6 months, or recurrent or metastatic cancer.
* Autoimmune diseases: such as lupus, rheumatoid arthritis, Crohn's disease, ulcerative colitis
* Active infectious diseases (eg. HIV/AIDS, hepatitis C)
* Any underlying medical condition which in the opinion of the investigator would prohibit the patient from providing informed consent
* Major surgery within three months prior to the index event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for enrollment include:
  1. Ischemic stroke within 24 hours of symptom onset.
  2. Transient Ischemic Attack (TIA) within 24 hours of symptom onset.
  3. Non-ischemic transient neurologic event (TNE) within 24 hours of onset.
  4. Normal controls that will be non-neurologic patients who are matched with the other ischemic stroke and TIA patients for age, race, gender and smoking plus one or more of the following vascular risk factors: diabetes, hypertension, atrial fibrillation, hyperlipidemia.
Sampling Method: Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2013-12; Primary Completion 2019-11 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Cardioembolic and large vessel stroke stiology | Up to 60 days.
  Determine the ability of ISCDX, a blood test, to differentiate between clinically diagnosed cardioembolic and large artery atherosclerotic ischemic stroke when hemorrhagic stroke is ruled out.
TIA differentiation from non ischemic events (TNE). | Up to 60 days.
  Determine the ability of TIADX, a blood test, to identify clinically diagnosed TIAs and differentiate these events from controls, which include TNEs. TNEs represent patients presenting with clinical symptoms similar to a TIA such as migraines, seizures and syncope, which are non-ischemic transient neurological events (TNE).

SECONDARY OUTCOMES:
Cryptogenic stroke | Up to 60 days.
  Determine the ability of ISCDX to categorize strokes of cryptogenic strokes, as either cardioembolic or large artery atherosclerotic when best practice clinical diagnostic testing cannot determine the cause, suggesting the best treatment pathway.
Atrial fibrillation and stroke | Up to 60 days.
  Determine the ability of ISCDX to further sub-classify strokes diagnosed as cardioembolic into those caused by atrial fibrillation and those not caused by atrial fibrillation, such as structural defects in the heart.
Stroke and TIA, differentiation | Up to 60 days.
  Determine the ability of the ISCDX and TIADX tests to differentiate between a TIA and an ischemic stroke, much in the manner that Acute Coronary Syndrome is now viewed as part of a spectrum of cardiovascular diseases.

OTHER OUTCOMES:
Development of point of care testing for ischemic stroke, transient ischemic attack (TIA), and transient neurological events (TNE). | Up to 60 days.
  Investigate the ability to translate the primary and secondary objectives into platforms that may be used in acute ischemic stroke evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Peacock, MD, Principal Investigator — Ischemia Care; Edward Jauch, MD, Principal Investigator — Medical University of South Carolina
Locations (22):
- United States (22):
  - Dignity Health Mercury San Juan, Sacramento, California
  - Zuckerberg San Francisco General Hospital (UCSF), San Francisco, California
  - University of California San Francisco Medical Center Hospital, San Francisco, California
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital - Beaumont Health System, Royal Oak, Michigan
  - Washington University, University Hospital in St Louis, St Louis, Missouri
  - The Stroke Center at Saint Barnabas Medical Center, Livingston, New Jersey
  - Montefiore Medical Center (University Hospital for Albert Einstein College of Medicine), The Bronx, New York
  - University of North Carolina Department of Neurology - Stroke Division, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital/ Ohio Health Research Institute, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Providence Health and Services, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - UT Health Department of Neurology, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams HP Jr, Bendixen BH, Kappelle LJ, Biller J, Love BB, Gordon DL, Marsh EE 3rd. Classification of subtype of acute ischemic stroke. Definitions for use in a multicenter clinical trial. TOAST. Trial of Org 10172 in Acute Stroke Treatment. Stroke. 1993 Jan;24(1):35-41. doi: 10.1161/01.str.24.1.35. PMID 7678184
- [Background] Ovbiagele B, Saver JL, Fredieu A, Suzuki S, Selco S, Rajajee V, McNair N, Razinia T, Kidwell CS. In-hospital initiation of secondary stroke prevention therapies yields high rates of adherence at follow-up. Stroke. 2004 Dec;35(12):2879-83. doi: 10.1161/01.STR.0000147967.49567.d6. Epub 2004 Oct 28. PMID 15514170
- [Background] Ionita CC, Xavier AR, Kirmani JF, Dash S, Divani AA, Qureshi AI. What proportion of stroke is not explained by classic risk factors? Prev Cardiol. 2005 Winter;8(1):41-6. doi: 10.1111/j.1520-037x.2005.3143.x. PMID 15722693
- [Background] Stead LG, Gilmore RM, Bellolio MF, Jain A, Rabinstein AA, Decker WW, Agarwal D, Brown RD Jr. Cardioembolic but not other stroke subtypes predict mortality independent of stroke severity at presentation. Stroke Res Treat. 2011;2011:281496. doi: 10.4061/2011/281496. Epub 2011 Oct 10. PMID 22007347
- [Background] Kamel et al. J Stroke Cerebrolvasc Dis; 2009 Nov-Dec;18(6):453-7. The risk of stroke recurrence is four times greater among prior stroke patients with newly detected AF.
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Furie KL, Kasner SE, Adams RJ, Albers GW, Bush RL, Fagan SC, Halperin JL, Johnston SC, Katzan I, Kernan WN, Mitchell PH, Ovbiagele B, Palesch YY, Sacco RL, Schwamm LH, Wassertheil-Smoller S, Turan TN, Wentworth D; American Heart Association Stroke Council, Council on Cardiovascular Nursing, Council on Clinical Cardiology, and Interdisciplinary Council on Quality of Care and Outcomes Research. Guidelines for the prevention of stroke in patients with stroke or transient ischemic attack: a guideline for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Jan;42(1):227-76. doi: 10.1161/STR.0b013e3181f7d043. Epub 2010 Oct 21. PMID 20966421
- [Background] Jickling GC, Xu H, Stamova B, Ander BP, Zhan X, Tian Y, Liu D, Turner RJ, Mesias M, Verro P, Khoury J, Jauch EC, Pancioli A, Broderick JP, Sharp FR. Signatures of cardioembolic and large-vessel ischemic stroke. Ann Neurol. 2010 Nov;68(5):681-92. doi: 10.1002/ana.22187. PMID 21031583
- [Background] Jickling GC, Zhan X, Stamova B, Ander BP, Tian Y, Liu D, Sison SM, Verro P, Johnston SC, Sharp FR. Ischemic transient neurological events identified by immune response to cerebral ischemia. Stroke. 2012 Apr;43(4):1006-12. doi: 10.1161/STROKEAHA.111.638577. Epub 2012 Feb 2. PMID 22308247
- [Background] Tang Y, Lu A, Aronow BJ, Sharp FR. Blood genomic responses differ after stroke, seizures, hypoglycemia, and hypoxia: blood genomic fingerprints of disease. Ann Neurol. 2001 Dec;50(6):699-707. doi: 10.1002/ana.10042. PMID 11761467
- [Background] Tang Y, Xu H, Du X, Lit L, Walker W, Lu A, Ran R, Gregg JP, Reilly M, Pancioli A, Khoury JC, Sauerbeck LR, Carrozzella JA, Spilker J, Clark J, Wagner KR, Jauch EC, Chang DJ, Verro P, Broderick JP, Sharp FR. Gene expression in blood changes rapidly in neutrophils and monocytes after ischemic stroke in humans: a microarray study. J Cereb Blood Flow Metab. 2006 Aug;26(8):1089-102. doi: 10.1038/sj.jcbfm.9600264. Epub 2006 Jan 4. PMID 16395289
- [Background] Xu H, Tang Y, Liu DZ, Ran R, Ander BP, Apperson M, Liu XS, Khoury JC, Gregg JP, Pancioli A, Jauch EC, Wagner KR, Verro P, Broderick JP, Sharp FR. Gene expression in peripheral blood differs after cardioembolic compared with large-vessel atherosclerotic stroke: biomarkers for the etiology of ischemic stroke. J Cereb Blood Flow Metab. 2008 Jul;28(7):1320-8. doi: 10.1038/jcbfm.2008.22. Epub 2008 Apr 2. PMID 18382470
- [Background] Stamova B, Xu H, Jickling G, Bushnell C, Tian Y, Ander BP, Zhan X, Liu D, Turner R, Adamczyk P, Khoury JC, Pancioli A, Jauch E, Broderick JP, Sharp FR. Gene expression profiling of blood for the prediction of ischemic stroke. Stroke. 2010 Oct;41(10):2171-7. doi: 10.1161/STROKEAHA.110.588335. Epub 2010 Aug 26. PMID 20798371
- [Background] Jickling GC, Stamova B, Ander BP, Zhan X, Tian Y, Liu D, Xu H, Johnston SC, Verro P, Sharp FR. Profiles of lacunar and nonlacunar stroke. Ann Neurol. 2011 Sep;70(3):477-85. doi: 10.1002/ana.22497. Epub 2011 Jul 27. PMID 21796664
- [Background] Zhan X, Jickling GC, Tian Y, Stamova B, Xu H, Ander BP, Turner RJ, Mesias M, Verro P, Bushnell C, Johnston SC, Sharp FR. Transient ischemic attacks characterized by RNA profiles in blood. Neurology. 2011 Nov 8;77(19):1718-24. doi: 10.1212/WNL.0b013e318236eee6. Epub 2011 Oct 12. PMID 21998319
- [Background] Jickling GC, Stamova B, Ander BP, Zhan X, Liu D, Sison SM, Verro P, Sharp FR. Prediction of cardioembolic, arterial, and lacunar causes of cryptogenic stroke by gene expression and infarct location. Stroke. 2012 Aug;43(8):2036-41. doi: 10.1161/STROKEAHA.111.648725. Epub 2012 May 24. PMID 22627989
- [Background] Jauch EC, Barreto AD, Broderick JP, Char DM, Cucchiara BL, Devlin TG, Haddock AJ, Hicks WJ, Hiestand BC, Jickling GC, June J, Liebeskind DS, Lowenkopf TJ, Miller JB, O'Neill J, Schoonover TL, Sharp FR, Peacock WF. Biomarkers of Acute Stroke Etiology (BASE) Study Methodology. Transl Stroke Res. 2017 May 5;8(5):424-8. doi: 10.1007/s12975-017-0537-3. Online ahead of print. PMID 28477280